CLINICAL TRIAL: NCT05718518
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and PK of ASC11/RTV Tablets and Study to Evaluate the Effects of Food on the PK of ASC11/RTV Tablets in Healthy Subjects
Brief Title: Study to Evaluate Safety, Tolerability, PK and the Food Effect on PK of ASC11/RTV Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC11-101
Record Dates: First submitted 2023-01-06; First posted 2023-02-08 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Healthy; COVID-19
Keywords: COVID-19; ASC11; 3CL-pro
MeSH Terms: conditions — COVID-19 | interventions — Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASC11 tablets (Experimental): Part 1: Subjects will receive ASC11 tablets on single ascending doses with proposed dose levels of ASC11 tablets: 100mg (cohort 1), 200 mg (cohort 2), 400mg (cohort 3) and 800 mg (cohort 4).
  Part 2: Subjects will receive ASC11tablets 100 to 300 mg (including 3 cohorts) and ASC11 tablets 300 mg(cohort 4) twice daily (BID) for 5 consecutive days and receive a single dose in the early morning of Day 6.
  Part 3: Subjects will be randomized to receive ASC11 tablets two single 200 mg or 300 mg doses (fed or fasted)
  Interventions: Drug: ASC11 tablets
- RTV tablets (Experimental): Part 1: Subjects will receive RTV tablets on 100 mg (cohort 1-4). Part 2: Subjects will receive RTV tablets 100 mg (including 3 cohorts) twice daily (BID) for 5 consecutive days and receive a single dose in the early morning of Day 6.
  Part 3: Subjects will be randomized to receive two single 100 mg doses (fed or fasted)
  Interventions: Drug: RTV tablets
- Placebo (Placebo Comparator): Part 1 and 2: Subjects will be randomized to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC11 tablets — Part 1: Subjects will receive ASC11 tablets on single ascending doses with proposed dose levels of ASC11 tablets: 100mg (cohort 1), 200 mg (cohort 2), 400mg (cohort 3) and 800 mg (cohort 4).
  Part 2: Subjects will receive ASC11tablets 100 to 300 mg (including 3 cohorts) and ASC11 tablets 300 mg(cohort 4) twice daily (BID) for 5 consecutive days and receive a single dose in the early morning of Day 6.
  Part 3: Subjects will be randomized to receive ASC11 tablets two single 200 mg or 300 mg doses (fed or fasted)
  Arms: ASC11 tablets
Drug: Placebo — Part 1 and 2: Subjects will be randomized to receive placebo.
  Arms: Placebo
Drug: RTV tablets — Part 1: Subjects will receive RTV tablets on 100 mg (cohort 1-4). Part 2: Subjects will receive RTV tablets 100 mg (including 3 cohorts) twice daily (BID) for 5 consecutive days and receive a single dose in the early morning of Day 6.
  Part 3: Subjects will be randomized to receive two single 100 mg doses (fed or fasted)
  Arms: RTV tablets

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I clinical study evaluating the safety, tolerability, and pharmacokinetics of ASC11 plus ritonavir tablets in healthy subjects and an open-label, cross-over study evaluating the effect of food on the pharmacokinetics of ASC11 plus ritonavir tablets

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged 18-60 years (including boundary values)
* If a woman has no planned pregnancy within 6 months after signing the informed consent, and is willing to use effective contraception (e.g. condom, uterine cap, non-hormonal intrauterine device [IUD]) for at least 3 months from the first administration of the study intervention to the last administration of the study intervention; Or not fertile (e.g. surgical sterilization [bilateral oophorectomy, tubal ligation, or hysterectomy] or natural sterilization [continuous > 12 months without menstruation])
* If male, agree to use effective contraception throughout the study intervention and for at least 3 months after the last dose of the study intervention, and do not donate sperm.
* General good health based on history, physical examination (screening and check-in assessment), vital signs and other screening assessments.
* Able to understand the research content, comply with the research protocol, and voluntarily sign the informed consent.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with acute or chronic diseases, including but not limited to cardiovascular, digestive, respiratory, urinary, nervous, endocrine, immune, musculoskeletal, and skin conditions, were judged by the investigator.
* Any previous or existing hematological disorders or disorders, major liver disease, family history of bleeding/platelet disease.
* Previous or existing cancer (other than basal cell carcinoma or squamous cell carcinoma of the skin), or hygrosis.
* Have an autoimmune disease, immunosuppression, or any form of immune deficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) of ASC11 relative to placebo | From screening through study completion, up to 14 days
  To evaluate the safety and tolerability of ASC11 tablets combined with Ritonavir tablets in healthy subjects given single and multiple dose increments.

SECONDARY OUTCOMES:
Title Pharmacokinetics (PK) parameter of ASC11 tablets combined with Ritonavir tablets in Plasma: AUC 0-inf | From screening through study completion, up to 14 days
  Area under the concentration-time curve from the time of dosing extrapolated to time infinity
Title -Pharmacokinetics (PK) parameter of ASC11 tablets combined with Ritonavir tablets in Plasma: Cmax | From screening through study completion, up to 14 days
  Maximum concentration
Pharmacokinetics (PK) parameter of ASC11 tablets combined with Ritonavir tablets in Plasma: Tmax | From screening through study completion, up to 14 days
  Time to Maximum Observed Plasma Concentration
Pharmacokinetics (PK) parameter of ASC11 tablets combined with Ritonavir tablets in Plasma: AUC 0-t | From screening through study completion, up to 14 days
  Area under the concentration-time curve from the time of dosing to the last measurable concentration
Pharmacokinetics (PK) parameter of ASC11 tablets combined with Ritonavir tablets in Plasma: T1/2 | From screening through study completion, up to 14 days
  Elimination half-life
Pharmacokinetics (PK) parameter of ASC11 tablets combined with Ritonavir tablets in Plasma: CL/F | From screening through study completion, up to 14 days
  Apparent total systemic clearance
Pharmacokinetics (PK) parameter of ASC11 tablets combined with Ritonavir tablets in Plasma: Vz/F | From screening through study completion, up to 14 days
  Apparent volume of distribution during the terminal elimination phase
Pharmacokinetics (PK) parameter of ASC11 tablets in Urine: CLR | From screening through study completion, up to 14 days
  Renal clearance

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China